CLINICAL TRIAL: NCT02312206
Title: A Phase 3, Randomized, Multicenter, Double-Blind, Placebo-Controlled, 2-Arm, Efficacy and Safety Study of NEOD001 Plus Standard of Care Versus Placebo Plus Standard of Care in Subjects With Light Chain (AL) Amyloidosis
Brief Title: The VITAL Amyloidosis Study, a Global Phase 3, Efficacy and Safety Study of NEOD001 in Patients With AL Amyloidosis
Acronym: VITAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The VITAL study was terminated due to futility analysis
Sponsor: Prothena Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEOD001-CL002
Record Dates: First submitted 2014-12-02; First posted 2014-12-09 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Primary Systemic (AL) Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — birtamimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NEOD001 (Experimental): 24 mg/kg (maximum dose of 2500 mg) of NEOD001 administered once every 28 days.
  Interventions: Drug: NEOD001
- Placebo (Placebo Comparator): Placebo will be administered as a 250 mL bag of normal saline once every 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NEOD001 — NEOD001, is a humanized immunoglobulin G1 monoclonal antibody, which specifically targets misfolded light chain aggregates and amyloid deposits. NEOD001 is proposed for use to target the misfolded light chain protein in subjects with AL amyloidosis.
  Arms: NEOD001
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, international, randomized, double-blind, placebo-controlled, two-arm efficacy and safety study in subjects newly diagnosed with AL amyloidosis. Subjects will remain on-study until study completion, which will occur when all primary endpoint events (all-cause mortality or cardiac hospitalizations) have been reached.

DETAILED DESCRIPTION:
This is a multi-center, international, randomized, double-blind, placebo-controlled, two-arm efficacy and safety study in subjects newly diagnosed with AL amyloidosis. Approximately 236 subjects will be enrolled in ~60 centers, with approximately 118 subjects per arm.

This is an event driven trial, therefore subjects will remain on-study until study completion, which will occur when all primary endpoint events (all-cause mortality or cardiac hospitalizations) have been reached. All subjects who discontinue will be followed until the last event is adjudicated. The estimated overall study duration is approximately 42 months, including the enrollment and treatment periods

Study drug will be administered once every 28 days as a 60-120 minute IV infusion.

First-line chemotherapy must be a bortezomib-containing regimen, with bortezomib administered weekly. The number of cycles of first-line chemotherapy that are administered are at the discretion of the Investigator, and subsequent chemotherapy regimens may be prescribed as per standard of care at the Investigator's discretion.

An independent Data Monitoring Committee (DMC) will review data on a regular basis.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years
2. Newly diagnosed, AL amyloidosis treatment naïve
3. Bone marrow consistent with plasma cell dyscrasia
4. Confirmed diagnosis of AL amyloidosis
5. Cardiac involvement
6. Planned first-line chemotherapy contains a proteasome-inhibiting agent administered weekly
7. Adequate bone marrow reserve, hepatic and renal function

Key Exclusion Criteria:

1. Non-AL amyloidosis
2. Meets diagnostic criteria for symptomatic multiple myeloma
3. Subject is eligible for and plans to undergo ASCT
4. History of Grade ≥ 3 infusion-associated AEs or hypersensitivity to another monoclonal antibody, or known hypersensitivity to diphenhydramine or acetaminophen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-02; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (79):
- United States (32):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - Stanford Cancer Institute (SCI), Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Radiant Research Northwestern University, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in Saint Louis, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Columbia University - College of Physicians & Surgeons, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina Chapel Hill Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic - Main Campus, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburg - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas; MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Froedtert & Medical College of Wisconsin, Cancer Center-Froedtert Hospital, Milwaukee, Wisconsin
- Australia (3):
  - Eastern Health (Box Hill Hospital), Box Hill
  - Amyloidosis Clinic Cnr Darcy Road and Bridge St. Westmead, Sydney
  - The University of Queensland-Princess Alexandra Hospital (PAH), Woolloongabba
- Universitatsklinik fur Innere Medizin 1 Kinische Abteilung fur Onkologie Aligemeines Krankenhaus - Universitatskliniken, Vienna, Austria
- Belgium (3):
  - ZNA Stuivenberg, Antwerp
  - ULB Hopital Erasme, Brussels
  - UZ Gasthuisberg, Leuven
- Canada (4):
  - University of Calgary-Southern Alberta Cancer Research Institute, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Research Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Rigshospitalet, Copenhagen, Denmark
- France (8):
  - Hopital de la Cote de Nacre Avenue, Caen
  - Hopital Henri Mondor, Créteil
  - CHU Dijon - Hopital du Bocage, Dijon
  - Hôpital Dupuytren - CHU Limoges, Limoges
  - Hôpital Pitié-Salpêtrière, Paris
  - Hopitaux Lyon Sud, Pierre-Bénite
  - Service d'Hermatologie CHU de Poitiers, Poitiers
  - CHU Rennes, Service de Medecine Interne, Rennes
- Germany (4):
  - Charite-Universitatsmedizin, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitatsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Universitatsklinikum Heidelberg, Heidelberg
- Greece (2):
  - Alexandra General Hospital of Athens, Athens
  - University Hospital of Patras, Pátrai
- Israel (4):
  - Hadassah University Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - Policlinico S.Orsola Malpighi, Unita' Operativa di Ematologia, Bologna
  - Policlinica San Matteo, Pavia
  - Azienda Ospedaliera Sant'Andrea, U.O.S., Rome
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- MTZ Clinical Research Sp. z o.o., Warsaw, Poland
- Spain (5):
  - Clínica Universidad de Navarra, Pamplona, Nevarra
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro - Maiadahonda, Madrid
- United Kingdom (6):
  - University Hospitals Birmingham NHS Foundation Trust - Queen Elizabeth Hospital, Birmingham
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology and Oncology Centre, Bristol
  - Leicester Royal Infirmary, Leicester
  - The Royal Free London NHS Foundation Trust-The Royal Free Hospital, London
  - NNUH NHS Foundation Trust - Norfolk and Norwich University Hospital, Norwich
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Gertz MA, Cohen AD, Comenzo RL, Kastritis E, Landau HJ, Libby EN, Liedtke M, Sanchorawala V, Schonland S, Wechalekar A, Zonder JA, Palladini G, Walling J, Guthrie S, Nie C, Karp C, Jin Y, Kinney GG, Merlini G. Birtamimab plus standard of care in light-chain amyloidosis: the phase 3 randomized placebo-controlled VITAL trial. Blood. 2023 Oct 5;142(14):1208-1218. doi: 10.1182/blood.2022019406. PMID 37366170

RESULTS

PARTICIPANT FLOW:
Groups:
- NEOD001 (24 mg/kg) + Standard of Care: NEOD001, 24 mg/kg IV every 28 days on top of standard of care until completion of 156 primary endpoints
- Placebo + Standard of Care: Placebo, 0.9% Saline IV every 28 days on top of standard of care until completion of 156 primary endpoints
Period: Overall Study
Arm/Group | NEOD001 (24 mg/kg) + Standard of Care | Placebo + Standard of Care
Started | 130 | 130
Informed Consent Obtained | 130 | 130
Completed | 0 | 0
Not Completed | 130 | 130
Not completed — Adverse Event | 3 | 6
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Physician Decision | 7 | 6
Not completed — Death | 31 | 36
Not completed — Study Terminated by Sponsor | 81 | 74
Not completed — Patient transferred to hospice | 0 | 1
Not completed — Subject missed three consecutive treatment visits | 0 | 1
Not completed — Patient progression and institution of a new therapy | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants
Groups:
- NEOD001 (24 mg/kg) + Standard of Care: NEOD001, 24 mg/kg IV every 4 weeks on top of Standard of Care
- Placebo + Standard of Care: Placebo 0.9% Saline IV every 4 weeks on top of Standard of Care
- Total: Total of all reporting groups
Arm/Group | NEOD001 (24 mg/kg) + Standard of Care | Placebo + Standard of Care | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 70 | 139
  >=65 years | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.69 (9.478) | 63.24 (9.708) | 63.46 (9.578)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 40 | 88
  Male | 82 | 90 | 172
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 118 | 120 | 238
  Black Or African American | 9 | 3 | 12
  Race not Reported | 1 | 5 | 6
  Asian | 2 | 2 | 4
  Hispanic Or Latino | 2 | 2 | 4
  Not Hispanic Or Latino | 116 | 122 | 238
  Ethnicity Not Reported | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Time to Composite of All-cause Mortality or Cardiac Hospitalization
Description: Time to all-cause mortality death occurring after the first infusion of study drug or cardiac hospitalization as adjudicated by the CEC occurring at least 91 days after first infusion of study drug through last subject last visit, whichever came first
Time Frame: Randomization until the date of death or cardiac hospitalization, up to 32 months
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | NEOD001 (24 mg/kg) + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 130 | 130
Participants
  Number of Subjects Who Died or Experienced Cardiac Hospitalization | 56 | 62
  Number of Subjects Censored | 74 | 68
Statistical Analysis 1: Comparison: NEOD001 (24 mg/kg) + Standard of Care vs Placebo + Standard of Care; Test type: Superiority; p = 0.3028, Log Rank; Hazard Ratio (HR) = 0.826, 95% CI 2-sided [0.5735 to 1.1889]

ADVERSE EVENTS:
Time Frame: Initiation of study drug through the last study visit or up to 30 days after last dose, whichever is later
Description: AE that newly appears, increases in frequency, or worsens in severity following initiation of study drug and through the last study visit or up to 30 days after date of last dose, whichever is later up to 32 months
Arm/Group | NEOD001 (24 mg/kg) + Standard of Care | Placebo + Standard of Care
All-Cause Mortality (participants affected / at risk) | 41/130 | 42/130
Serious Adverse Events (participants affected / at risk) | 88/130 | 91/130
Other Adverse Events (participants affected / at risk) | 124/130 | 125/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NEOD001 (24 mg/kg) + Standard of Care (N=130) | Placebo + Standard of Care (N=130)
Cardiac failure (Cardiac disorders) | 17 | 28
Cardiac failure congestive (Cardiac disorders) | 15 | 9
Cardiac arrest (Cardiac disorders) | 9 | 10
Atrial fibrillation (Cardiac disorders) | 6 | 6
Cardiac failure acute (Cardiac disorders) | 5 | 5
Ventricular tachycardia (Cardiac disorders) | 2 | 5
Acute myocardial infarction (Cardiac disorders) | 3 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 2 | 0
Cardiac amyloidosis (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 13 | 12
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 4 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0
Bronchitis (Infections and infestations) | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Injection site cellulitis (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pasteurella infection (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Ileus (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 3
Colitis (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 4 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 1
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Cell death (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 11 | 7
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 0 | 2
Brain injury (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Bell's palsy (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 7 | 9
Renal failure (Renal and urinary disorders) | 2 | 4
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Gastrointestinal disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sudden death (General disorders) | 1 | 3
Death (General disorders) | 1 | 2
Generalised oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 2
Malaise (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 1
Non-cardiac Chest pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 6
Orthostatic hypotension (Vascular disorders) | 2 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acquired factor VIII deficiency (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic haematoma (Hepatobiliary disorders) | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Myocardial necrosis marker increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Mania (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amyloidosis (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NEOD001 (24 mg/kg) + Standard of Care (N=130) | Placebo + Standard of Care (N=130)
Constipation (Gastrointestinal disorders) | 54 | 55
Diarrhoea (Gastrointestinal disorders) | 51 | 54
Nausea (Gastrointestinal disorders) | 56 | 43
Vomiting (Gastrointestinal disorders) | 25 | 20
Abdominal distension (Gastrointestinal disorders) | 15 | 15
Abdominal pain (Gastrointestinal disorders) | 14 | 14
Stomatitis (Gastrointestinal disorders) | 7 | 8
Abdominal pain upper (Gastrointestinal disorders) | 6 | 8
Dry mouth (Gastrointestinal disorders) | 6 | 7
Dysphagia (Gastrointestinal disorders) | 7 | 5
Oedema peripheral (General disorders) | 55 | 56
Fatigue (General disorders) | 57 | 52
Pyrexia (General disorders) | 12 | 11
Asthenia (General disorders) | 8 | 8
Chills (General disorders) | 9 | 4
Dizziness (Nervous system disorders) | 25 | 38
Neuropathy peripheral (Nervous system disorders) | 29 | 18
Headache (Nervous system disorders) | 17 | 16
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 13
Paraesthesia (Nervous system disorders) | 10 | 13
Dysgeusia (Nervous system disorders) | 8 | 9
Syncope (Nervous system disorders) | 7 | 11
Hypoaesthesia (Nervous system disorders) | 8 | 4
Upper respiratory tract infection (Infections and infestations) | 23 | 25
Urinary tract infection (Infections and infestations) | 14 | 6
Nasopharyngitis (Infections and infestations) | 8 | 10
Pneumonia (Infections and infestations) | 10 | 8
Respiratory tract infection (Infections and infestations) | 1 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 27
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 26 | 26
Decreased appetite (Metabolism and nutrition disorders) | 26 | 20
Hyponatraemia (Metabolism and nutrition disorders) | 16 | 17
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 4
Weight decreased (Investigations) | 19 | 16
Blood creatinine increased (Investigations) | 22 | 11
Aspartate aminotransferase increased (Investigations) | 11 | 8
Weight increased (Investigations) | 6 | 11
Platelet count decreased (Investigations) | 4 | 10
Alanine aminotransferase increased (Investigations) | 5 | 8
Lymphocyte count decreased (Investigations) | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Insomnia (Psychiatric disorders) | 39 | 30
Depression (Psychiatric disorders) | 11 | 7
Anxiety (Psychiatric disorders) | 11 | 3
Rash (Skin and subcutaneous tissue disorders) | 14 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 14
Ecchymosis (Skin and subcutaneous tissue disorders) | 7 | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 7
Hypotension (Vascular disorders) | 19 | 29
Orthostatic hypotension (Vascular disorders) | 9 | 13
Fall (Injury, poisoning and procedural complications) | 14 | 11
Contusion (Injury, poisoning and procedural complications) | 8 | 9
Anaemia (Blood and lymphatic system disorders) | 20 | 27
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 8
Lymphopenia (Blood and lymphatic system disorders) | 6 | 7
Atrial fibrillation (Cardiac disorders) | 8 | 10
Cardiac failure (Cardiac disorders) | 10 | 6
Palpitations (Cardiac disorders) | 3 | 11
Acute kidney injury (Renal and urinary disorders) | 8 | 4
Chronic kidney disease (Renal and urinary disorders) | 7 | 6
Haematuria (Renal and urinary disorders) | 2 | 7
Dry eye (Eye disorders) | 4 | 7
Vision blurred (Eye disorders) | 8 | 1
Blood alkaline phosphatase increased (Investigations) | 12 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI, institution and the sponsor have agreed that the PI and institution may publish or disclose study results from their site after the earlier of (a) publication of the complete multicenter study results or (b) 18 months after database lock for the multicenter study. The sponsor has at least 45 days to review a proposed publication and may request deletion of confidential information and up to 60 days additional delay to obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT02312206/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT02312206/SAP_001.pdf